CLINICAL TRIAL: NCT04578392
Title: MeSenteric SpAring Versus High Ligation Ileocolic Resection for the Prevention of REcurrent Crohn's DiseaSe (SPARES)
Acronym: SPARES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Amy Lightner, Associate Professor of Surgery in the Department of Colon and Rectal Surgery at Cleveland Clinic, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-139
Record Dates: First submitted 2020-10-01; First posted 2020-10-08 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Crohn Disease
Keywords: ileocolic resection; Crohn's disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Intervention Model Description: Patients will be randomized according to post-operative recurrence risk to either a high ligation of ileocolic artery or mesenteric sparing ileocolic resection for terminal ileal Crohn's disease.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high ligation of ileocolic artery (Active Comparator): Randomized control trial of two operative techniques Operative approach of a high ligation of ileocolic artery as compared to mesenteric sparing for a primary ileocolic resection
  Interventions: Procedure: high ligation of ileocolic artery; Procedure: mesenteric sparing
- mesenteric sparing for a primary ileocolic resection (Active Comparator): Randomized control trial of two operative techniques Operative approach of a high ligation of ileocolic artery as compared to mesenteric sparing for a primary ileocolic resection
  Interventions: Procedure: high ligation of ileocolic artery; Procedure: mesenteric sparing

INTERVENTIONS:
Procedure: high ligation of ileocolic artery — Patients will be randomized according to post-operative recurrence risk to surgery to high ligation or mesenteric sparing
Procedure: mesenteric sparing — Patients will be randomized according to post-operative recurrence risk to surgery to high ligation or mesenteric sparing

SUMMARY:
Study description - Patients will be randomized according to post-operative recurrence risk to either a high ligation of ileocolic artery or mesenteric sparing ileocolic resection for terminal ileal Crohn's disease. The primary endpoint 6-month endoscopic recurrence.

Endpoints - Primary endpoint; 6 months Secondary endpoints at 1 and 5 years post ileocecal resection

Study population - Adult Crohn's disease patients with medically refractory terminal ileal Crohn's disease undergoing a primary ileocecal resection.

Study sites - Multicenter international study

Description of study intervention - Randomized control trial of two operative techniques Operative approach of a high ligation of ileocolic artery as compared to mesenteric sparing for a primary ileocolic resection

Participate duration - 5 years

DETAILED DESCRIPTION:
There is increasing evidence to suggest that the mesentery may play an active role in the pathophysiology of Crohn's disease. There is significant clinical, endoscopic, and surgical recurrence of disease following ileocolic resection at the site of the anastomosis. The study is seeking to understand if the mesentery plays a role in recurrence following ileocolic resection.

Crohn's disease (CD) is a chronic inflammatory disease of the intestinal tract with an unknown etiology and an unknown cure. The characteristic transmural inflammation can progress to refractory inflammatory disease, stricturing disease, and fistulizing disease - all potential indications for surgery when medical management has been exhausted. An important tenant to remember is that surgery is not curative but is rather an adjunct to maximal medical therapy.

One third of patients with Crohn's disease (CD) will require a major abdominal resection within 5 years of their diagnosis, and two-thirds will ultimately require operative management at least once during the course of their disease.

Unfortunately, surgery for Crohn's disease (CD) is not curative and disease recurrence is common with 62% having endoscopic recurrence at six months, and 80% and 30% of patients having endoscopic and clinical recurrence, respectively, at one year. A third of these patients will require a reoperation at 10 years and up to 80% will require an additional operation by 15 years.This undoubtedly leads to an increased probability of malabsorption syndrome and decreased quality of life.

A significant volume of research has been conducted in attempt to determine how to prevent postoperative recurrence of CD following an ileocolic resection. Some studies have focused on the timing of resuming postoperative medical therapy. Others have looked at surgical technique at the time of ileocolic resection including anatomic configuration of the anastomosis and performing a stapled versus handsewn anastomosis. Various configurations include a side to side anastomosis, end to end, and Kono-S anastomosis. A randomized clinical trial compared a side to side versus an end to end, and found endoscopic recurrence rates were similar in the two groups (42.5% versus 37.9%) at a mean follow up of 11.9 months. A later multi-institution international trial of the Kono S anastomosis determined that the anastomosis was associated with a decreased surgical recurrence rate as compared to conventional anastomoses; 5 and 10 year surgical recurrence-free survival was 98.6%.15 Several Cochrane Database reviews have reported no difference in a stapled versus handsewn anastomosis for an ileocolic resection. Therefore, other than the potential decreased recurrence with the Kono-S anastomosis, no other surgical techniques have altered the postoperative recurrence rate of CD following an ileocolic resection.

Interestingly there is recent evidence to suggest that CD may be a disease of the mesentery rather than just the mucosa of the bowel alone. In CD, the transmural inflammation facilitates increased bacterial translocation into the creeping fat. These translocating antigens and activate adipocytes which are cells than have complex metabolic and immunologic functions. Additionally, it is thought that functional abnormalities in the mesenteric structures exert an inflammatory effect: the secretion of adipokines that have endocrine functions contribute to immunomodulation through a response to afferent signals, neuropeptides, and functional cytokines; mesenteric nerves are involved in the pathogenesis through neuropeptides; and lymphatics in the mesentery may obstruct, remodel, and impair contraction, contributing to the irregularly thickened mesentery seen in CD. Interestingly, the interaction between neuropeptides, adipokines, and vascular and lymphatic endothelia leads to adipose tissue remodeling. This makes the mesentery an active participant in CD, seemingly as much as the bowel itself. However, the mesentery is typically spared, or left in situ, during resection for CD, unlike resections for adenocarinocma of the colon. In adenocarcinoma, a 'high ligation' is performed, where the feeding vessel is taken at its origin in order to take sufficient mesentery and lymph nodes with the colon specimen. However, in operations for CD, the mesentery is spared and typically taken close to the bowel wall despite enlarged lymph nodes and thickened diseased mesentery. A high ligation of the ileocolic artery in order to sample an increased volume of mesentery and lymph nodes to prevent postoperative CD has never been evaluated in a randomized control trial. A recent retrospective study comparing surgical recurrence following a mesenteric sparing versus mesenteric resection approach with ileocecal resection found cumulative reoperation rates were significantly lower in the mesenteric resection group (40% versus 2.9%; p=0.003).

The endoscopic recurrence of CD typically precedes clinical symptoms, and the severity of lesions can predict the subsequent symptomatic course of the disease. Over a four year follow-up period, 100% of patients with severe endoscopic recurrence (Rutgeerts score of i2-i4) developed symptomatic recurrence compared to only 9% of patients with a low score (i0-i1). With such a high rate of endoscopic recurrence, it is thought that post-surgical evaluation should be performed at six months rather than one year when considering adequate early treatment.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18-65 years of age.
* Isolated ileocolic Crohn's disease of <30 cm in length
* Concurrent therapies with corticosteroids, 5-ASA drugs, thiopurines, MTX, antibiotics, anti-TNF, vedolizumab, ustekinumab therapy are permitted.
* Ability to comply with protocol
* Competent and able to provide written informed consent
* Medically refractory disease or inability to tolerate ongoing medical therapy

Exclusion Criteria:Inability to give informed consent.

* Patients less than 18 years of age
* Patients undergoing repeat ileocolic resection
* Patients with concurrent disease in other locations (e.g. proximal stricturing of the small bowel, fistulizing disease to the sigmoid colon) requiring an additional intervention in the operating room beyond an ileocolic resection.
* Patients with >30 cm of terminal ileal disease
* Patients who are undergoing an ileal resection only (NOT ileocecal) because the disease spares the distal most aspect of ileum and ileocecal valve
* Patient whose anastomosis is diverted intra-operatively with a loop or end ileostomy
* Clinically significant medical conditions within the six months before surgery: e.g. myocardial infarction, active angina, congestive heart failure or other conditions that would, in the opinion of the investigators, compromise the safety of the patient.
* Specific exclusions; Evidence of hepatitis B, C, or HIV
* History of cancer including melanoma (with the exception of localized skin cancers)
* Emergent indication for an operation
* Pregnant or breast feeding.
* History of clinically significant auto-immunity (other than Crohn's disease) or any previous example of fat-directed autoimmunity
* Inability to follow up at respective sites for the primary endpoint

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Estimated)
Dates: Start 2020-07-28 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Endoscopic recurrence based on Rutgeert scoring at the time of colonoscopy | 6 months
  Endoscopic recurrence is define as a Rutgeert score >2 at the time of colonoscopy The score is attributed directly, by selecting the appropriate degree - 5 degrees, from i0 (lowest) to i4 highest, with single-choice selection menu. Rutgeerts score is only be used for evaluation of post-surgical recurrences at ileocolic anastomosis level.

SECONDARY OUTCOMES:
Clinical Recurrence - Crohn's Disease Activity Index (CDAI) | 6 months, 1 year
  Clinical Recurrence is defined as an increase in CDAI >100 or CDAI >150
  This tool used to quantify the symptoms of patients with Crohn's disease in order to define response or remission of disease. Remission of Crohn's disease is defined as CDAI below 150. Severe disease was defined as a value of greater than 450. Most major research studies on medications in Crohn's disease define response as a fall of the CDAI of greater than 70 points. (score ranges form 0 to over 600, the higher the score, the higher the disease state)
Endoscopic Recurrence - Rutgeert score | 1 year
  Endoscopic recurrence is define as a score >2 at the time of colonoscopy The score is attributed directly, by selecting the appropriate degree - 5 degrees, from i0 (lowest) to i4 highest, with single-choice selection menu. Rutgeerts score is only be used for evaluation of post-surgical recurrences at ileocolic anastomosis level.
Surgical Recurrence | 1 and 5 years
  Surgical recurrence is define as need for repeat ileocolic resection due to recurrence at anastomotic site

CONTACTS AND LOCATIONS:
Overall Officials: Amy Lightner, MD, Principal Investigator — The Cleveland Clinic
Locations (7):
- United States (4):
  - Cedars-Sinai Hospital System, Los Angeles, California
  - Stanford University School of Medicine, Stanford, California
  - Cleveland Clinic Florida, Weston, Florida
  - Cleveland Clinic, Cleveland, Ohio
- Mt. Sinai, Toronto, Ontario, Canada
- Humanitas, Rozzano, Milano, Italy
- St Mark's Hospital and Academic Institution, Harrow, Middlesex, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bernell O, Lapidus A, Hellers G. Risk factors for surgery and postoperative recurrence in Crohn's disease. Ann Surg. 2000 Jan;231(1):38-45. doi: 10.1097/00000658-200001000-00006. PMID 10636100
- [Background] Bouguen G, Peyrin-Biroulet L. Surgery for adult Crohn's disease: what is the actual risk? Gut. 2011 Sep;60(9):1178-81. doi: 10.1136/gut.2010.234617. Epub 2011 May 24. No abstract available. PMID 21610273
- [Background] Peyrin-Biroulet L, Oussalah A, Williet N, Pillot C, Bresler L, Bigard MA. Impact of azathioprine and tumour necrosis factor antagonists on the need for surgery in newly diagnosed Crohn's disease. Gut. 2011 Jul;60(7):930-6. doi: 10.1136/gut.2010.227884. Epub 2011 Jan 12. PMID 21228429
- [Background] Canin-Endres J, Salky B, Gattorno F, Edye M. Laparoscopically assisted intestinal resection in 88 patients with Crohn's disease. Surg Endosc. 1999 Jun;13(6):595-9. doi: 10.1007/s004649901049. PMID 10347299
- [Background] Mekhjian HS, Switz DM, Watts HD, Deren JJ, Katon RM, Beman FM. National Cooperative Crohn's Disease Study: factors determining recurrence of Crohn's disease after surgery. Gastroenterology. 1979 Oct;77(4 Pt 2):907-13. No abstract available. PMID 467942
- [Background] Lewis RT, Maron DJ. Efficacy and complications of surgery for Crohn's disease. Gastroenterol Hepatol (N Y). 2010 Sep;6(9):587-96. PMID 21088749
- [Background] Lazarev M, Ullman T, Schraut WH, Kip KE, Saul M, Regueiro M. Small bowel resection rates in Crohn's disease and the indication for surgery over time: experience from a large tertiary care center. Inflamm Bowel Dis. 2010 May;16(5):830-5. doi: 10.1002/ibd.21118. PMID 19798731
- [Background] Orlando A, Mocciaro F, Renna S, Scimeca D, Rispo A, Lia Scribano M, Testa A, Aratari A, Bossa F, Tambasco R, Angelucci E, Onali S, Cappello M, Fries W, D'Inca R, Martinato M, Castiglione F, Papi C, Annese V, Gionchetti P, Rizzello F, Vernia P, Biancone L, Kohn A, Cottone M. Early post-operative endoscopic recurrence in Crohn's disease patients: data from an Italian Group for the study of inflammatory bowel disease (IG-IBD) study on a large prospective multicenter cohort. J Crohns Colitis. 2014 Oct;8(10):1217-21. doi: 10.1016/j.crohns.2014.02.010. Epub 2014 Mar 11. PMID 24630485
- [Background] Olaison G, Smedh K, Sjodahl R. Natural course of Crohn's disease after ileocolic resection: endoscopically visualised ileal ulcers preceding symptoms. Gut. 1992 Mar;33(3):331-5. doi: 10.1136/gut.33.3.331. PMID 1568651
- [Background] Rutgeerts PJ. From aphthous ulcer to full-blown Crohn's disease. Dig Dis. 2011;29(2):211-4. doi: 10.1159/000323922. Epub 2011 Jul 5. PMID 21734386
- [Background] Michelassi F, Balestracci T, Chappell R, Block GE. Primary and recurrent Crohn's disease. Experience with 1379 patients. Ann Surg. 1991 Sep;214(3):230-8; discussion 238-40. doi: 10.1097/00000658-199109000-00006. PMID 1929605
- [Background] Rutgeerts P. Strategies in the prevention of post-operative recurrence in Crohn's disease. Best Pract Res Clin Gastroenterol. 2003 Feb;17(1):63-73. doi: 10.1053/bega.2002.0358. PMID 12617883
- [Background] McLeod RS, Wolff BG, Ross S, Parkes R, McKenzie M; Investigators of the CAST Trial. Recurrence of Crohn's disease after ileocolic resection is not affected by anastomotic type: results of a multicenter, randomized, controlled trial. Dis Colon Rectum. 2009 May;52(5):919-27. doi: 10.1007/DCR.0b013e3181a4fa58. PMID 19502857
- [Background] Kono T, Fichera A, Maeda K, Sakai Y, Ohge H, Krane M, Katsuno H, Fujiya M. Kono-S Anastomosis for Surgical Prophylaxis of Anastomotic Recurrence in Crohn's Disease: an International Multicenter Study. J Gastrointest Surg. 2016 Apr;20(4):783-90. doi: 10.1007/s11605-015-3061-3. Epub 2015 Dec 22. PMID 26696531
- [Background] Neutzling CB, Lustosa SA, Proenca IM, da Silva EM, Matos D. Stapled versus handsewn methods for colorectal anastomosis surgery. Cochrane Database Syst Rev. 2012 Feb 15;2012(2):CD003144. doi: 10.1002/14651858.CD003144.pub2. PMID 22336786
- [Background] Choy PY, Bissett IP, Docherty JG, Parry BR, Merrie A, Fitzgerald A. Stapled versus handsewn methods for ileocolic anastomoses. Cochrane Database Syst Rev. 2011 Sep 7;(9):CD004320. doi: 10.1002/14651858.CD004320.pub3. PMID 21901690
- [Background] Kredel L, Batra A, Siegmund B. Role of fat and adipokines in intestinal inflammation. Curr Opin Gastroenterol. 2014 Nov;30(6):559-65. doi: 10.1097/MOG.0000000000000116. PMID 25188546
- [Background] Li Y, Zhu W, Zuo L, Shen B. The Role of the Mesentery in Crohn's Disease: The Contributions of Nerves, Vessels, Lymphatics, and Fat to the Pathogenesis and Disease Course. Inflamm Bowel Dis. 2016 Jun;22(6):1483-95. doi: 10.1097/MIB.0000000000000791. PMID 27167572
- [Background] Coffey CJ, Kiernan MG, Sahebally SM, Jarrar A, Burke JP, Kiely PA, Shen B, Waldron D, Peirce C, Moloney M, Skelly M, Tibbitts P, Hidayat H, Faul PN, Healy V, O'Leary PD, Walsh LG, Dockery P, O'Connell RP, Martin ST, Shanahan F, Fiocchi C, Dunne CP. Inclusion of the Mesentery in Ileocolic Resection for Crohn's Disease is Associated With Reduced Surgical Recurrence. J Crohns Colitis. 2018 Nov 9;12(10):1139-1150. doi: 10.1093/ecco-jcc/jjx187. PMID 29309546
- [Background] Rutgeerts P, Geboes K, Vantrappen G, Beyls J, Kerremans R, Hiele M. Predictability of the postoperative course of Crohn's disease. Gastroenterology. 1990 Oct;99(4):956-63. doi: 10.1016/0016-5085(90)90613-6. PMID 2394349
- [Result] Caprilli R, Gassull MA, Escher JC, Moser G, Munkholm P, Forbes A, Hommes DW, Lochs H, Angelucci E, Cocco A, Vucelic B, Hildebrand H, Kolacek S, Riis L, Lukas M, de Franchis R, Hamilton M, Jantschek G, Michetti P, O'Morain C, Anwar MM, Freitas JL, Mouzas IA, Baert F, Mitchell R, Hawkey CJ; European Crohn's and Colitis Organisation. European evidence based consensus on the diagnosis and management of Crohn's disease: special situations. Gut. 2006 Mar;55 Suppl 1(Suppl 1):i36-58. doi: 10.1136/gut.2005.081950c. PMID 16481630